CLINICAL TRIAL: NCT02590029
Title: Psychosocial Support for Acute Hospital Pain and Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Garland, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00085446
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Mindfulness; Suggestion

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Mindfulness (Experimental): 15 minute mindfulness session
  Interventions: Behavioral: Mindfulness
- Suggestion (Experimental): 15 minute therapeutic suggestion session
  Interventions: Behavioral: Suggestion
- Psychoeducation (Active Comparator): 15 minute psychoeducation session
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness — The 15 minute mindfulness session is a scripted mindfulness exercise that incorporates mindfulness principles of intentionally paying attention to present-moment experience in a non-judgmental fashion.
  Arms: Mindfulness
Behavioral: Suggestion — The 15 minute suggestion session is a scripted suggestion exercise that incorporates imagery and suggestions for changes in cognition, emotion, and body sensations.
  Arms: Suggestion
Behavioral: Psychoeducation — The 15 minute psychoeducation session is a supportive session in which behavioral coping strategies for pain management are discussed.
  Arms: Psychoeducation

SUMMARY:
The purpose of this randomized study is to determine the impact of three different types of psychosocial support delivered by social workers to patients reporting uncontrolled pain during a hospital stay. This study will examine the differential effects of brief mindfulness training, therapeutic suggestion, and psychoeducation for patients reporting uncontrolled pain.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking males or females 18 or older within the University of Utah Hospital system reporting "intolerable pain" or "inadequate pain control" on the Clinically Aligned Pain Assessment Tool (CAPA; Donaldson & Chapman, 2013).

Exclusion Criteria:

* Altered mental status due to delirium, psychosis, or pharmacological sedation as determined by clinical assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity (numeric rating scale) | Immediately prior to and following intervention
  0-10 scale
Pain unpleasantness (numeric rating scale) | Immediately prior to and following intervention
  0-10 scale

SECONDARY OUTCOMES:
Use of opioid analgesics | 24 hours prior to and following intervention
  The total amount of opioid analgesic use will be computed during the 24 hours prior to and following intervention. Opioid dose will be standardized and calculated using conventional morphine daily equivalent equianalgesic conversion tables.
Anxiety (numeric rating scale) | Immediately prior to and following intervention
  0-10 scale
Relaxation (numeric rating scale) | Immediately prior to and following intervention
  0-10 scale
Desire for opioids (numeric rating scale) | Immediately prior to and following intervention
  0-10 scale
Positive body sensations (numeric rating scale) | Immediately prior to and following intervention
  0-10 scale
Use of non-opioid analgesics (NSAID) | Within 24 hours prior to and following intervention
  The total amount of opioid analgesic use will be computed during the 24 hours prior to and following intervention. NSAID dose will be standardized and calculated using conventional NSAID equianalgesic conversion tables.

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Garland, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Donaldson, G., & Chapman, C.R. (2013). Pain management is more than just a number. University of Utah Health/Department of Anesthesiology. Salt Lake City, Utah: Department of Anesthesiology.
- [Derived] Garland EL, Baker AK, Larsen P, Riquino MR, Priddy SE, Thomas E, Hanley AW, Galbraith P, Wanner N, Nakamura Y. Randomized Controlled Trial of Brief Mindfulness Training and Hypnotic Suggestion for Acute Pain Relief in the Hospital Setting. J Gen Intern Med. 2017 Oct;32(10):1106-1113. doi: 10.1007/s11606-017-4116-9. Epub 2017 Jul 12. PMID 28702870